CLINICAL TRIAL: NCT02009072
Title: Comparison Between Sutureless and Glue Free Versus Sutured Limbal Conjunctival Autograft in Primary Pterygium Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaaban Elwan (Other)
Collaborators: Minia University (Other)
Responsible Party: Sponsor-Investigator, Shaaban Elwan, Assisstent professor of ophthalmology, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pterygium Surgery
Record Dates: First submitted 2013-12-02; First posted 2013-12-11 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Pterygium
Keywords: Pterygium surgery; Sutureless glue free conjunctival autograft; Amniotic membrane graft.
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sutured limbal conjunctival autograft (Experimental): Sutured limbal conjunctival autograft was done for patients of group 2 after pterygium excision
  Interventions: Procedure: Sutured limbal conjunctival autograft
- Suturless and glue free Limbal conjuctival autograft (Experimental): Sutureless and glue free Limbal conjunctival autograft was done for patients of group 1 after pterygium excision
  Interventions: Procedure: Sutureless and glue free limbal conjunctival autograft

INTERVENTIONS:
Procedure: Sutureless and glue free limbal conjunctival autograft — Simple pterygium excision under local anesthesia was performed then closure of the bare sclera by sutureless and glue free conjunctival autograft in 50 eyes of 50 patients (group 1)
  Other Names: Sutureless and glue free LCAG
  Arms: Suturless and glue free Limbal conjuctival autograft
Procedure: Sutured limbal conjunctival autograft — Simple pterygium excision under local anesthesia was performed then closure of the bare sclera by sutured limbal conjunctival autograft in 100 eyes of 100 patients (group 2).
  Other Names: Sutured LCAG
  Arms: Sutured limbal conjunctival autograft

SUMMARY:
Pterygium is a common ocular pathology facing ophthalmologists that has varied surgical management techniques and high rate of post-operative recurrence. The investigators aim was to compare and evaluate the safety and efficacy outcomes of those two surgical procedures in management of primary pterygium.

DETAILED DESCRIPTION:
Design: Prospective randomized clinical trial comparative study. Setting: Department of ophthalmology, Al-Minia University Faculty of medicine, Egypt.

Methods: The study included 150 eyes of 150 patients of primary pterygium. Twenty four to 74 years of age (mean 49 ± 12 years). Simple excision under local anesthesia was performed then closure of the bare sclera by sutureless and glue free conjunctival autograft in 50 eyes of 50 patients (group 1), versus sutured free conjunctival autograft in 100 eyes of 100 patients (group 2).

ELIGIBILITY:
Inclusion Criteria:

Patients complaining of primary pterygium with eye redness. Patients with pterygium threatening the visual axis.

Exclusion Criteria:

All cases not completed the follow up period for two years. Atrophic pterygium, pseudopterygium or double head pterygium.

Ages: 24 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Recurrence Rate | 24 months
  The main postoperative primary outcomes measure the recurrence rate which was defined as fibrovascular proliferation invading the cornea more than 1.5 mm at the site of previously excised pterygium.

SECONDARY OUTCOMES:
Postoperative signs and symptoms | Third postoperative day,then weekly for one month
  The secondary outcomes measure, postoperative pain, foreign body sensation, photophobia, hyperemia and chemosis.
Overall patient satisfaction | Third post-operative week
  Overall satisfaction with the procedure 3 weeks post-operatively was recorded as four grades 0= unsatisfied, 1= low satisfaction, 2= moderate satisfaction and 3= highly satisfied, the data were collected as mean scores and recorded. The two groups were compared for overall satisfaction.
Complications | 24 months
  Complications was recorded including, persistent epithelial defect, dellen, inclusion cyst, pyogenic granuloma, conjunctival edema, corneal scleral necrosis, infective scleritis, keratitis and endophthalmitis.

OTHER OUTCOMES:
Operative time | Intraoperative
  Calculation of operative time for each patient procedure
Gain in uncorrected visual acuity (UCVA) | First post-operative month
  Gain in uncorrected visual acuity (UCVA) for each patient from the base line measurement

CONTACTS AND LOCATIONS:
Overall Officials: Shaaban A Elwan, Assist Prof Ophth, Principal Investigator — Ophthalmology Dep., Al-Minya University Hospitals, Al-Minya, Egypt
Locations (1):
- Shaaban A Elwan, Al Minyā, Egypt